CLINICAL TRIAL: NCT03022331
Title: VCRC Longitudinal Protocol for Aortitis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Peter Merkel, Chief, Division of Rheumatology Professor of Medicine and Epidemiology, University of Pennsylvania
Other Study IDs: VCRC5507; U54AR057319 (NIH)
Record Dates: First submitted 2016-12-20; First posted 2017-01-16 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Aortitis
Keywords: Idiopathic aortitis; Isolated aortitis; Vasculitis
MeSH Terms: conditions — Aortitis; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples, including genetic information (DNA), will be collected from patients with aortitis in this study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational

SUMMARY:
The term 'aortitis' refers to inflammation of the aorta. Aortitis is known to occur in a variety of vasculitides and connective tissue diseases, such as giant cell arteritis (GCA), Takayasu arteritis (TAK), rheumatoid arthritis, and spondyloarthropathies, among others. This study will establish a longitudinal cohort for these diseases.

DETAILED DESCRIPTION:
This study will develop a longitudinal cohort of patients with different types of aortitis to systematically study the natural history, optimal treatments, and outcomes in this group of diseases. This will provide a resource for future studies and for identification of new biomarkers of aortitis for purposes of diagnosis, disease activity measurement, disease damage assessment, determination of disease states, and evaluation of treatment response.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if they meet one of the following criteria:

1. Previous or current microscopic evidence of aortitis (active or healed) on surgical specimen obtained during aortic resection
2. Previous or current radiographic aortitis that could include circumferential aortic wall thickening of at least 3mm on CT or MRI or increased PET FDG uptake in the aorta at values equal to or greater than the liver, in absence of an alternative explanation for the radiographic findings.

Exclusion

1. Subjects already enrolled in one of the other VCRC longitudinal cohorts: 5502, 5503, 5504, 5505, and 5506.
2. Inability of participants (or their guardians in the case of children) to give informed consent and to sign the consent form.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 250 patients with aortitis will be enrolled into the VCRC longitudinal observational cohort study and followed for up to ten years. The study will be conducted at major vasculitis centers in North America, utilizing the Clinical and Translational Science Center (CTSC) at each site.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Phenotypic correlates of genotype | 5 years
  Using longitudinally collected phenotypic data, this project aims to define the natural history (i.e. biochemical evidence of systemic inflammation, and systemic symptoms) of different types of phenotypes of aortitis and related disorders in patients using serum and genetic information collected through specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Milman, MD, MSc, Principal Investigator — University of Ottawa; Peter A Merkel, MD, MPH, Study Director — University of Pennsylvania
Locations (10):
- United States (7):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (3):
  - University British Columbia/Mary Pack Arthritis Centre, Vancouver, British Columbia
  - St. Joseph's Healthcare, Hamilton, Ontario
  - University of Toronto, Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- See also: Related Info — http://www.rarediseasesnetwork.org/vcrc